CLINICAL TRIAL: NCT00802529
Title: Effectiveness of Transtympanic Steroids in Unilateral Ménière's Disease: a Randomised Controlled Double-Blind Trial
Brief Title: Transtympanic Gentamicin vs. Steroids in Refractory Meniere's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO1135
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Meniere's Disease
Keywords: Meniere's disease; transtympanic steroids; Randomised controlled trial
MeSH Terms: conditions — Meniere Disease | interventions — Methylprednisolone; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid (Methylprednisolone) (Experimental): Steroid (Methylprednisolone)
  Interventions: Drug: Methylprednisolone
- Gentamicin (Active Comparator): Gentamicin
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Methylprednisolone — 2 transtympanic injections at interval of two weeks.
  Arms: Steroid (Methylprednisolone)
Drug: Gentamicin — 2 transtympanic injections at an interval of two weeks. If there is significant hearing loss before second injection, it will be replaced by normal saline in double blinded fashion.
  Arms: Gentamicin

SUMMARY:
This trial aims to compare transtympanic steroids against the standard treatment (transtympanic gentamicin) in refractory unilateral Meniere's disease.

DETAILED DESCRIPTION:
Meniere's disease is characterised by episodic spontaneous vertigo attacks with hearing loss, ringing sounds and fullness in the ear. In one out of five patients, standard first line medical treatment is not effective in controlling vertigo attacks. For these incapacitated patients, gentamicin injections through the ear drum is a well established minimally invasive treatment. Major surgery of the balance organs or nerve, risking complete hearing loss, CSF leak, meningeal infections, are rarely performed nowadays. Gentamicn is very effective in controlling vertigo and acts by chemical ablation of end organs. As hearing and balance organs are entwined around each other, gentamicin treatment does not come without the risk of hearing loss. In fact, meta-analysis shows hearing deterioration in 13% to 35% percent of gentamicin treated patients. On the other hand, steroids are drug of choice for autoimmune inner ear disease and commonly used for sudden hearing loss. They are non toxic drugs without any known side effects during local treatment in ear. We will compare the two in this randomised, double blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral Ménière's disease (definite or probable, according to Committee on Hearing and Equilibrium guidelines, 1995) with hearing loss and presenting with recurrent vertigo, not responding to medical treatment for at least 6 months will be included. There should be normal, age appropriate hearing in the contralateral ear.

Exclusion Criteria:

* Patients with Ménière's disease in later stages (not having vertigo attacks).
* Age: patients older than 70 years at the start of the trial.
* Severe disability (e.g. neurological, orthopaedic, cardiovascular) or serious concurrent illness that might interfere with treatment or follow up.
* Active additional neuro-otological disorders that may mimic Ménière's disease (e.g. vestibular migraine, vertebro-basilar TIAs, acoustic neuroma) and thus will make the objective follow up difficult.
* Concurrent ear pathology that may interfere with transtympanic treatment (e.g. active middle ear disease).
* Family history of unexplained deafness (possibility of genetic susceptibility to gentamicin toxicity).
* History of known adverse/allergic reaction to steroids or gentamicin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo M Bronstein, PhD, FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial college Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Sjogren J, Fransson PA, Magnusson M, Karlberg M, Tjernstrom F. Acute unilateral vestibulopathy and corticosteroid treatment - A randomized placebo-controlled double-blind trial. J Vestib Res. 2025 Mar;35(2):91-101. doi: 10.1177/09574271241307649. Epub 2024 Dec 18. PMID 39973595
- [Derived] Patel M, Agarwal K, Arshad Q, Hariri M, Rea P, Seemungal BM, Golding JF, Harcourt JP, Bronstein AM. Intratympanic methylprednisolone versus gentamicin in patients with unilateral Meniere's disease: a randomised, double-blind, comparative effectiveness trial. Lancet. 2016 Dec 3;388(10061):2753-2762. doi: 10.1016/S0140-6736(16)31461-1. Epub 2016 Nov 17. PMID 27865535

RESULTS

PARTICIPANT FLOW:
Groups:
- Steroid (Methylprednisolone): Methylprednisolone: 2 transtympanic injections at interval of two weeks. Each injection was 62.5mg/ml.
- Gentamicin: Gentamicin: 2 transtympanic injections at an interval of two weeks. If there is significant hearing loss before second injection, it will be replaced by normal saline in double blinded fashion.Each injection was 40mg/ml.
Period: Overall Study
Arm/Group | Steroid (Methylprednisolone) | Gentamicin
Started | 30 | 30
Completed | 30 (2 patients crossed-over to gentamicin after steroids failed to control vertigo (as per protocol).) | 29
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid (Methylprednisolone) | Gentamicin | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (10.2) | 53.3 (10.8) | 52.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 20 | 15 | 35
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Vertigo Attacks
Description: The number of vertigo attacks between 18-24months follow-up were taken retrospectively during a face-to-face appointment at 24 months follow-up and compared to 6 month pre-enrollment baseline (as per Committee on Hearing and Equilibrium guidelines).
Time Frame: 6month pre-enrollment baseline, 18-24 months after initial treatment
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: Vertigo Attacks
Arm/Group | Steroid (Methylprednisolone) | Gentamicin
Number analyzed (Participants) | 30 | 29
Vertigo Attacks
  Baseline | 16.4 (12.45) | 19.93 (16.7)
  18-24months | 1.6 (3.4) | 2.5 (5.8)
Statistical Analysis 1: Comparison: Steroid (Methylprednisolone) vs Gentamicin; Test type: Superiority or Other; p = 0.271, ANOVA — P-value for Drug x Time interaction; Time: 2 degrees of freedom (Baseline vs 18-24 months) Drug: 2 degrees of freedom (Gentamicin vs steroid)

2. Secondary Outcome: Change in Hearing
Description: Hearing was measured as ipsilesional pure-tone threshold at Baseline, 1month, 2months, 6months, 12month, 18months and 24 months follow-up. Hearing level was taken as the average threshold across 0.5, 1, 2 and 3KHz.
Time Frame: Baseline, 1,2,6,12,18 and 24months after initial treatment
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Steroid (Methylprednisolone) | Gentamicin
Number analyzed (Participants) | 30 | 29
dB
  Baseline | 53.25 (21.17) | 51.5 (11.29)
  1month | 49.29 (22.23) | 52.18 (15.77)
  2months | 49.83 (22.31) | 48.99 (16.9)
  6months | 46.67 (23.29) | 45.48 (17.7)
  12months | 47.02 (23.96) | 47.34 (19.2)
  18months | 48.44 (22.1) | 44.82 (18.8)
  24months | 46.9 (24.0) | 49.1 (18.1)
Statistical Analysis 1: Comparison: Steroid (Methylprednisolone) vs Gentamicin; Test type: Superiority or Other; p = 0.964, ANOVA — P-value for Drug x Time interaction; Time: 6 degrees of freedom (Baseline, 1, 2, 6, 12, 18 and 24 months) Drug: 2 degrees of freedom (Gentamicin vs steroid)

3. Secondary Outcome: Change in Speech Discrimination
Description: Speech discrimination was measured at Baseline, 1month, 2months, 6months, 12month and 24 months follow-up.
  Speech discrimination was assessed by means of ipsilesional suprathreshold word recognition (%). Arthur Boothroyd's isophonemic word lists (AB wordlists, Guymark, Southampton) comprising sets of 10 words were played to the ipsilesional ear at the low-frequency pure-tone threshold of 0·5, 1 and 2 kHz +30dB with masking sound in the contralesional ear if necessary. The formula for masking level was: low-frequency pure-tone threshold in ipsilesional ear - bone conduction mean threshold (0·5, 1 and 2KHz) in contralesional ear - 40dB. Speech loudness and masking were rounded to the nearest 5dB. Step increments and decrements of 10dB for speech loudness and masking were used to attain the maximum speech discrimination score.
Time Frame: Baseline, 1,2,6,12 and 24months after initial treatment
Measure: Mean (Standard Deviation); unit: Percentage correct
Arm/Group | Steroid (Methylprednisolone) | Gentamicin
Number analyzed (Participants) | 30 | 29
Percentage correct
  Baseline | 64.97 (29.28) | 72.10 (21.67)
  1month | 71.78 (26.48) | 69.43 (22.94)
  2months | 76.10 (24.43) | 74.31 (23.4)
  6months | 75.63 (26.39) | 76.35 (25.92)
  12months | 73.43 (27.16) | 71.58 (24.69)
  24months | 76.32 (29.36) | 64.99 (30.75)
Statistical Analysis 1: Comparison: Steroid (Methylprednisolone) vs Gentamicin; Test type: Superiority or Other; p = 0.128, ANOVA — P-value for Drug x Time interaction; Time: 5 degrees of freedom (Baseline, 1, 2, 6, 12 and 24 months) Drug: 2 degrees of freedom (Gentamicin vs steroid)

ADVERSE EVENTS:
Arm/Group | Steroid (Methylprednisolone) | Gentamicin
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 3/30 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid (Methylprednisolone) (N=30) | Gentamicin (N=32)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Retinoschisis (Eye disorders) | 1 (1) | 0 (0)
Scwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cist (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes